CLINICAL TRIAL: NCT00729729
Title: Phase 4, Three Way Cross-over, Pharmacokinetic Study for PCA Derivate Formulations in Healthy Subjects
Brief Title: Pharmacokinetic Study for PCA Derivate Formulations
Acronym: PCA 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Gadi Lalazar MD, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: PCA pharmacokinetics 1
Record Dates: First submitted 2008-08-03; First posted 2008-08-07 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Comparative; bioavailability; of PCA; formulations
MeSH Terms: interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: PCA
- 2 (Experimental): Slow release PCA derivative
  Interventions: Drug: PCA
- 3 (Experimental): Slow release PCA derivative higher dose
  Interventions: Drug: PCA

INTERVENTIONS:
Drug: PCA — Placebo tablet, once
  Arms: 1
Drug: PCA — PO, 700mg, once
  Arms: 2
Drug: PCA — PO, 1000mg, once
  Arms: 3

SUMMARY:
A comparative bioavailability study of PCA slow release versus immediate release formulations, after a single dose to fasting healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the informed consent process culminating with written informed consent by the subject.
* Males
* Age 18-45 years
* Abstinence from alcohol for 1 week prior to the study
* Non smoking
* BMI > 19 and < 30
* No history or evidence of significant

  * cardiovascular,
  * hepatic,
  * renal,
  * hematopoietic,
  * gastrointestinal disease,
  * endocrine,
  * metabolic,
  * psychiatric
  * psychological disorders
* Normal physical examination
* Within +/- 10% of normal values in laboratory examinations

Exclusion Criteria:

* Subjects who suffer from a current medical condition.
* Subjects who smoke.
* Subjects who drink > 20 grams of alcohol per day.
* Subjects who take prescription medication.
* Subjects with an abnormality in screening blood tests
* Known sensitivity to any ingredients in the study drug

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PCA derivate blood levels | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel